CLINICAL TRIAL: NCT00178061
Title: Treatment of Primary Mood Disorders in the Comorbidly Ill
Brief Title: Effects of Comorbid Personality Disorder on the Treatment of Bipolar I Disorder
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Pittsburgh (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 970843-0109; 970843-0109
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Last update posted 2013-06-25 (Estimated); Status verified 2013-06

CONDITIONS: Bipolar I Disorder; Borderline Personality Disorder
MeSH Terms: conditions — Borderline Personality Disorder

INTERVENTIONS:
Behavioral: Interpersonal Social Rhythm Therapy (IPSRT)

SUMMARY:
This study will examine the impact of comorbid personality disorder on the outcome of treatment among patients with bipolar I disorder.

DETAILED DESCRIPTION:
The major aim of this proposal is to examine the impact of comorbid personality disorder on the outcome of treatment among patients with bipolar I disorder.

The specific aims are to create a research and supervisory team and to identify potential moderators of treatment response and mediators of outcome over the course of treatment.

Members of the team will meet weekly to begin a treatment development process for enhancing Interpersonal Social Rhythm Therapy (IPSRT) for these patients. Additional assessment measures will be utilized to examine the proposed mediators and moderators of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Bipolar I Disorder with Comorbid Borderline Personality Disorder, currently manic or depressed

Exclusion Criteria:

* Unstable Medical illness

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 13
Dates: Start 1997-08; Study Completion 2002-08

PRIMARY OUTCOMES:
Hamilton Rating Scale for Depression (HRSD-25)

SECONDARY OUTCOMES:
Raskin Severity of Depression and Mania Scales

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Frank, Principal Investigator — University of Pittsburgh
Locations (1):
- Western Psychiatric Institute and Clinic, Pittsburgh, Pennsylvania, United States